CLINICAL TRIAL: NCT02339519
Title: A Comparison of Supraglottic Airway Devices; Lma Classic, Lma Fastrach and Lma Supreme; a Prospective, Randomized, Clinical Trial of Efficacy, Safety and Complications
Brief Title: A Comparison of Supraglottic Airway Devices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GK4
Record Dates: First submitted 2015-01-03; First posted 2015-01-15 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Airway Management
Keywords: Laryngeal Masks

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- group LMA supreme (Active Comparator): Patients who received Laryngeal Mask Airway; LMA supreme
  Interventions: Device: LMA SUPREME
- group LMA classic (Active Comparator): Patients who received Laryngeal Mask Airway; LMA classic
  Interventions: Device: LMA CLASSIC
- group Fastrach (Active Comparator): Patients who received Laryngeal Mask Airway; LMA fastrach
  Interventions: Device: LMA FASTRACH

INTERVENTIONS:
Device: LMA CLASSIC — Classic LMA consists of a mask with a surrounding inflatable bag compatible to the shape of the hypopharynx and a tube that has a 30° angle with a mask.
  Arms: group LMA classic
Device: LMA FASTRACH — Fastrach LMA has similar features to the LMA Classic, but it is designed to provide upper airway during intubation via blind intubation or fiberoptic assistance. It has a rigid handle that allows one-handed insertion, removal or adjustment.
  Arms: group Fastrach
Device: LMA SUPREME — Supreme LMA is a novel, sterile, single use, new generation supraglottic airway device which provides more rapid and higher volume gas passage through airway and can be inserted in a rapid and safe manner.
  Arms: group LMA supreme

SUMMARY:
This study aimed to compare the advantages and disadvantages of LMA Supreme, LMA Classic and LMA Fastrach regarding ease of insertion, repositioning, insertion time, effects on hemodynamic parameters, provision of adequate and safe airway, and oropharyngeal and systemic complications.

DETAILED DESCRIPTION:
As a result of studies regarding the provision of an airway which is less invasive than intubation but safer than mask to maintain patency of airway after anesthesia induction in brief surgical interventions, supraglottic airway devices have been introduced into practice. They are inserted to glottic entry via the oral route and can be used in emergent conditions where tracheal intubation and mask anesthesia are challenging.

Classic LMA was first introduced by Archie Brain, MD in 1988, and consists of a mask with a surrounding inflatable bag compatible to the shape of the hypopharynx and a tube that has a 30° angle with a mask.

Fastrach LMA ( LMA Fastrach: LMA North America. Inc. San Diego. CA) was first introduced in 1997 and has similar features to the LMA Classic, but it is designed to provide upper airway during intubation via blind intubation or fiberoptic assistance. It has a rigid handle that allows one-handed insertion, removal or adjustment.

Supreme LMA, first introduced in April, 2007, is a novel, sterile, single use, new generation supraglottic airway device which provides more rapid and higher volume gas passage through airway and can be inserted in a rapid and safe manner because of the advanced cuff and airway tube. The integrated gastric canal facilitates gastric aspiration.

Supraglottic airway devices seem to have advantages over each other in different aspects due to their distinct features. In literature, there are studies comparing various LMA types for different features. However, to best of our knowledge, there is no study comparing these 3 types of LMA regarding these parameter. This is the main point of difference of our study.

ELIGIBILITY:
Inclusion Criteria:

* normotensive patients with mouth aperture > 3 cm,
* thyromental distance > 6 cm,
* sternomental distance > 12.5 cm,
* body mass index < 35 kg m-2 were included in the study.

Exclusion Criteria:

* patients with ASA III-IV,
* those with a history of gastroesophageal reflux,
* pregnancy,
* cardiovascular and central nerve system disease,
* those with difficulty in cooperation,
* those undergoing intracranial, intraabdominal and Ear-nose-throat surgeries were excluded from study.

None of the methods changed after commencement of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Ease of insertion will be rated using a 4-point scale (4: success at the first attempt without tactile resistance; 3: success at the first attempt with tactile resistance; 2: success at the second attempt; 1: failure at the second attempt). | 1 month

SECONDARY OUTCOMES:
Composite measure of Hemodynamic parameters , change 20% from baseline in Mean Blood Pressure and Heart Rate | baseline and 1 month
Number of Participants with oropharyngeal ( edema, haemorragie, blood in sputum) and systemic complications (anaflactic reactions) | 1 month
Time to successful insertion time and effective airway [ time to observation of 3 consequtive correct End-Tidal CO2 (EtCO2 )waves after insertion ] defined as insertion time and was recorded. | 1 monyh
Measure if the inserted device failed to provide adequate ventilation, the device position was changed within the oral cavity, which was then defined as repositioning | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Erdal Komur, MD, Principal Investigator — Istanbul Umraniye Education and Research Hospital
Locations (1):
- Istanbul Umraniye Education and Research Hospital, Istanbul, Turkey, Turkey (Türkiye)

REFERENCES:
- [Background] Timmermann A, Cremer S, Heuer J, Braun U, Graf BM, Russo SG. [Laryngeal mask LMA Supreme. Application by medical personnel inexperienced in airway management]. Anaesthesist. 2008 Oct;57(10):970-5. doi: 10.1007/s00101-008-1425-8. German. PMID 18712321
- [Background] Seet E, Rajeev S, Firoz T, Yousaf F, Wong J, Wong DT, Chung F. Safety and efficacy of laryngeal mask airway Supreme versus laryngeal mask airway ProSeal: a randomized controlled trial. Eur J Anaesthesiol. 2010 Jul;27(7):602-7. doi: 10.1097/eja.0b013e32833679e3. PMID 20540172